CLINICAL TRIAL: NCT01642277
Title: The Effect of Short Term Solifenacin for Overactive Bladder on the Female Urinary Microbiome
Brief Title: Bacterial Genomic Sequencing in Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Alan J. Wolfe, Professor, Microbiology Immunology, Loyola University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 204195
Record Dates: First submitted 2012-07-03; First posted 2012-07-17 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-10

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; OAB; Urinary Tract Infection; UTI; Microbiome; Bacteria; Solifenacin; 16S rRNA sequence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Tract Infections | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women using Solifenacin for OAB treatment (Experimental): Solifenacin treated women: Women with OAB who are prescribed solifenacin
  Interventions: Drug: Solifenacin
- Control: Women without OAB (No Intervention): Women without OAB who are not prescribed solifenacin.

INTERVENTIONS:
Drug: Solifenacin — 5 mg for 4 weeks with option to increase to 10 mg for an additional 8 weeks
  Other Names: Vesicare
  Arms: Women using Solifenacin for OAB treatment

SUMMARY:
No one really knows what causes overactive bladder syndrome (OAB). Urinary tract infection (UTI)causes similar symptoms to OAB with the difference being the presence of bacteria, as evidenced by routine microbiology cultures. Recent work by the group on the genitourinary microbiome (GUM) has shown that female urine, even in the absence of culture evidence of bacteria does have evidence of bacterial DNA. Bacterial 16S rRNA can be isolated from urine and sequenced to identify bacterial species present in urine. From this the investigators can hypothesize that urinary bacteria contribute to urinary symptoms and that there is a difference in the bacterial communities in the urine of women who respond to Solifenacin, a drug used to treat OAB, versus those that do not.

DETAILED DESCRIPTION:
This is a prospective study with two groups: Women who have accepted a clinical recommendation for OAB treatment with solifenacin and a comparator (control) group of women unaffected by OAB. All women will have a baseline urine assessment with bacterial genome sequencing. Solifenacin treated patients will also have urine assessments with bacterial genomic sequencing at 4 and 12 weeks on treatment.

ELIGIBILITY:
Inclusion Criteria:

Controls: Women without bother from urinary symptoms will be screened for potential study participation using the pelvic floor distress inventory (PFDI). Women with negative urinary responses will be further screened for participation using the following eligibility criteria:

* no anticholinergic medications for bladder conditions,
* no antibiotic exposure in the past 4 weeks for any reason,
* no immunologic deficiency,
* no pelvic malignancy or pelvic radiation, and
* Untreated symptomatic POP > POP-Q Stage II.

OAB cohort: Women with bother from overactive bladder symptoms will be screened for potential study participation using the pelvic floor distress inventory (PFDI). Women with positive urinary responses for urge predominant symptoms will be further screened for participation using the following eligibility criteria:

* willing to take Solifenacin as treatment for OAB,
* no neurological disease known to affect the lower urinary tract,
* no current UTI (based on urine dipstick) or recurrent UTI,
* no antibiotic exposure in the past 4 weeks for any reason,
* no immunologic deficiency,
* no pelvic malignancy or pelvic radiation,
* untreated symptomatic POP > POP-Q Stage II,
* no contraindications to receiving Solifenacin.

Exclusion Criteria:

* Women who are of child-bearing potential who are pregnant, nursing, intending to become pregnant during the study or not practicing a reliable form of contraception are also excluded.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Wolffe, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago Health Sciences Division, Maywood, Illinois, United States

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Hartmann KE, McPheeters ML, Biller DH, Ward RM, McKoy JN, Jerome RN, Micucci SR, Meints L, Fisher JA, Scott TA, Slaughter JC, Blume JD. Treatment of overactive bladder in women. Evid Rep Technol Assess (Full Rep). 2009 Aug;(187):1-120, v. PMID 19947666
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] de Boer TA, Salvatore S, Cardozo L, Chapple C, Kelleher C, van Kerrebroeck P, Kirby MG, Koelbl H, Espuna-Pons M, Milsom I, Tubaro A, Wagg A, Vierhout ME. Pelvic organ prolapse and overactive bladder. Neurourol Urodyn. 2010;29(1):30-9. doi: 10.1002/nau.20858. PMID 20025017
- [Background] Sajadi KP, Vasavada SP. Overactive bladder after sling surgery. Curr Urol Rep. 2010 Nov;11(6):366-71. doi: 10.1007/s11934-010-0136-2. PMID 20803179
- [Background] Mostwin JL. Pathophysiology: the varieties of bladder overactivity. Urology. 2002 Nov;60(5 Suppl 1):22-6; discussion 27. doi: 10.1016/s0090-4295(02)01788-0. PMID 12493346
- [Background] Michel MC, Chapple CR. Basic mechanisms of urgency: roles and benefits of pharmacotherapy. World J Urol. 2009 Dec;27(6):705-9. doi: 10.1007/s00345-009-0446-5. PMID 19588154
- [Background] Ohtake A, Sato S, Sasamata M, Miyata K. The forefront for novel therapeutic agents based on the pathophysiology of lower urinary tract dysfunction: ameliorative effect of solifenacin succinate (Vesicare), a bladder-selective antimuscarinic agent, on overactive bladder symptoms, especially urgency episodes. J Pharmacol Sci. 2010;112(2):135-41. doi: 10.1254/jphs.09r13fm. Epub 2010 Feb 4. PMID 20134114
- [Background] Hoffstetter S, Leong FC. Solifenacin succinate for the treatment of overactive bladder. Expert Opin Drug Metab Toxicol. 2009 Mar;5(3):345-50. doi: 10.1517/17425250902762866. PMID 19331596
- [Background] Pelman RS, Capo JP Jr, Forero-Schwanhaeuser S. Solifenacin at 3 years: a review of efficacy and safety. Postgrad Med. 2008 Jul;120(2):85-91. doi: 10.3810/pgm.2008.07.1795. PMID 18654073
- [Background] Haab F, Cardozo L, Chapple C, Ridder AM; Solifenacin Study Group. Long-term open-label solifenacin treatment associated with persistence with therapy in patients with overactive bladder syndrome. Eur Urol. 2005 Mar;47(3):376-84. doi: 10.1016/j.eururo.2004.11.004. Epub 2005 Jan 5. PMID 15716204
- [Background] Santos JC, Telo ER. Solifenacin: scientific evidence in the treatment of overactive bladder. Arch Esp Urol. 2010 Apr;63(3):197-213. English, Spanish. PMID 20431184
- [Background] Oliver JD. The viable but nonculturable state in bacteria. J Microbiol. 2005 Feb;43 Spec No:93-100. PMID 15765062
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Derived] Thomas-White KJ, Hilt EE, Fok C, Pearce MM, Mueller ER, Kliethermes S, Jacobs K, Zilliox MJ, Brincat C, Price TK, Kuffel G, Schreckenberger P, Gai X, Brubaker L, Wolfe AJ. Incontinence medication response relates to the female urinary microbiota. Int Urogynecol J. 2016 May;27(5):723-33. doi: 10.1007/s00192-015-2847-x. Epub 2015 Sep 30. PMID 26423260
- [Derived] Pearce MM, Hilt EE, Rosenfeld AB, Zilliox MJ, Thomas-White K, Fok C, Kliethermes S, Schreckenberger PC, Brubaker L, Gai X, Wolfe AJ. The female urinary microbiome: a comparison of women with and without urgency urinary incontinence. mBio. 2014 Jul 8;5(4):e01283-14. doi: 10.1128/mBio.01283-14. PMID 25006228
- [Derived] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on July 16th, 2012 and ended on May 22nd, 2014 (i.e., 22.2 months). Participants were recruited during their outpatient appointments to the Urogynecology Clinic at Loyola University Medical Center (Maywood, IL) by a member of the research team.
Pre-assignment Details: This was a 12-week open label study with no randomization scheme. Following diagnosis, patients were administered 5 mg daily solifenacin. At the 4-week visit, if a participant's symptoms were adequately controlled (response), she continued at dose for the study duration. If a participant reported no improvement, the dose was increased to 10 mg.
Groups:
- Urinary Urge Incontinence: Seventy-four (n = 74) women received 5-10mg daily solifenacin for the treatment of urinary urge incontinence (UUI).
- Non-Urinary Urge Incontinence: Sixty (n = 60) women without UUI were evaluated at baseline only (week 0) in order to serve as a control cohort. These women never received study therapy (i.e., 5-10mg daily solifenacin).
Period: Overall Study
Arm/Group | Urinary Urge Incontinence | Non-Urinary Urge Incontinence
Started | 74 | 60
Completed | 50 | 60
Not Completed | 24 | 0
Not completed — Adverse Event | 10 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 11 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses includes the baseline information of individuals lacking primary outcome measurements (i.e., patients that withdrew for any reason n = 24).
Groups:
- Urinary Urge Incontinence: Seventy-four (n = 74) women received 5mg daily solifenacin (with an option to increase to 10mg daily solifenacin at 4 weeks) for the treatment of urinary urge incontinence (UUI).
- Total: Total of all reporting groups
Arm/Group | Urinary Urge Incontinence | Non-Urinary Urge Incontinence | Total
Number analyzed (Participants) | 74 | 60 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.5) | 49 (14.7) | 56.04 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 60 | 134
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 56 | 43 | 99
  Black | 13 | 12 | 25
  Asian | 0 | 1 | 1
  Hispanic | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 74 | 60 | 134
Body Mass Index [Median (Standard Deviation); unit: kg/m2] | 32.7 (8.4) | 27.9 (5.5) | 30.59 (7.61)
Vaginal Parity [Median (Inter-Quartile Range); unit: Births] | 2.00 [1.00 to 3.00] | 2.00 [0 to 2.75] | 2.00 [0.00 to 3.00]
Estrogen Status [Number; unit: participants]
  Negative | 7 | 32 | 39
  Positive | 65 | 26 | 91
  Unknown | 2 | 2 | 4
Diabetes [Number; unit: participants]
  No | 67 | 58 | 125
  Yes | 7 | 2 | 9
Hypertension [Number; unit: participants]
  No | 48 | 49 | 97
  Yes | 26 | 11 | 37
Coronary Artery Disease [Number; unit: participants]
  No | 65 | 59 | 124
  Yes | 9 | 1 | 10
Smoking [Number; unit: participants]
  Non-Smoker | 68 | 56 | 124
  Smoker | 6 | 4 | 10
Marital Status [Number; unit: participants]
  Married | 38 | 37 | 75
  Separated | 3 | 1 | 4
  Divorced | 9 | 6 | 15
  Widowed | 14 | 1 | 15
  Single | 10 | 15 | 25
Prior Treatment for OAB [Number; unit: participants]
  Prior Treatment | 37 | 0 | 37
  No prior treatment | 37 | 60 | 97
Sequencing Urotypes at Baseline [Number; unit: participants]
  Low biomass | 37 | 34 | 71
  Lactobacillus urotype | 15 | 16 | 31
  Diverse urotype | 8 | 4 | 12
  Gardnerella urotype | 8 | 4 | 12
  Other urotypes | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Genomic Sequencing
Description: Participants were classified into Low Biomass, Lactobacillus, Gardnerella, Diverse, and Other urotypes based on the bacterial DNA at baseline.
Time Frame: 12 weeks
Population: This was a completer analysis comprising participants who completed 12 weeks of treatment (n = 50).
Measure: Number; unit: participants
Groups:
- Urinary Urge Incontinence: Women who received 5-10mg daily solifenacin for the treatment of urinary urge incontinence (UUI).
Arm/Group | Urinary Urge Incontinence
Number analyzed (Participants) | 50
participants
  Low biomass | 25
  Lactobacillus urotype | 11
  Diverse urotype | 3
  Gardnerella urotype | 6
  Other urotypes | 3

2. Secondary Outcome: Assessment of Overactive Bladder Questionnaire (OABQ)
Description: The Overactive Bladder Questionnaire (OAB-q) was developed to assess symptom bother and the impact of overactive bladder (OAB) on health-related quality of life (HRQL). The instrument comprises 33 items. Response options for the symptom frequency and HRQL items are presented as 6-point Likert scales ranging from 'none of the time' to 'all of the time' for symptom frequency (and 'not at all' to 'a very great deal' for symptom bother). From these 33 items, six sub-scales are assessed separately: (1) OAB symptom severity, (2) Coping with OAB symptoms, (3) Concern for OAB symptoms, (4) Sleep as a function of OAB symptoms, (5) Social functioning as a consequence of OAB symptoms, and (6) Health related quality of life (HRQL) as a function of OAB symptoms. Each sub-scale score ranges from 0 to 100 (where higher scores indicate more severe OAB symptoms and lower scores indicate minimal symptom severity).
Time Frame: End of study (Week 12)
Population: Participants who received solifenacin were asked to complete the OABQ at 12 weeks in order to assess overactive bladder symptoms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Solifenacin Responder: Individuals with urinary urge incontinence who responded to solifenacin at 12 weeks
- Solifenacin Non-Responder: Individuals with urinary urge incontinence who did not respond to solifenacin at 12 weeks
Arm/Group | Solifenacin Responder | Solifenacin Non-Responder
Number analyzed (Participants) | 37 | 13
units on a scale
  Symptom Severity Score | 17.50 [7.50 to 32.50] | 37.50 [15.00 to 61.25]
  Coping Score | 92.50 [85.00 to 100.00] | 80.00 [46.25 to 95.00]
  Concern Score | 97.14 [85.71 to 100.00] | 82.86 [41.43 to 95.71]
  Sleep Score | 92.00 [76.00 to 100.00] | 84.00 [50.00 to 96.00]
  Social Score | 100.00 [98.00 to 100.00] | 96.00 [80.00 to 100.00]
  Health Related Quality of Life (HRQL) | 92.80 [86.00 to 99.20] | 76.00 [63.20 to 95.20]
Statistical Analysis 1: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For symptom-severity score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size and non-normal distributions of symptom severity scores. The null hypothesis is that there is no difference between the two groups in symptom severity, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) symptom severity than the other group; Test type: Superiority or Other; p = .052, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.94
Statistical Analysis 2: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For coping score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size, non-normal distributions, and outliers of coping scores. The null hypothesis is that there is no difference between the two groups in coping, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) coping than the other group; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 2.06
Statistical Analysis 3: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the concern score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size, non-normal distributions, and outlier of the concern scores. The null hypothesis is that there is no difference between the two groups in their concern, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) concern than the other group; Test type: Superiority or Other; p = .03, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 2.176
Statistical Analysis 4: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the sleep score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size, non-normal distributions, and outliers of sleep scores. The null hypothesis is that there is no difference between the two groups in sleep scores, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) sleep scores than the other group; Test type: Superiority or Other; p = .37, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 0.90
Statistical Analysis 5: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For social score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size, non-normal distributions, and outliers of social scores. The null hypothesis is that there is no difference between the two groups in social scores, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) social scores than the other group; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 2.02
Statistical Analysis 6: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the overall health related quality of life (HRQL) score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size, non-normal distributions, and outliers of HRQL scores. The null hypothesis is that there is no difference between the two groups in health related quality of life, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) health realted quality of life than the other group; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 2.03

3. Secondary Outcome: Assessment of Pelvic Floor Disease Inventory (PFDI) Questionnaire
Description: The PFDI comprises 46 items on a 4-point symptom severity scale ranging from 1 = "Not at all" to 4 = "Quite a bit". From these items, 13 separate sub-scales are reported: (1) Obstructive discomfort, (2) Irritation, (3) Stress resulting from urinal distress, (4) A general sub-scale for pelvic organ prolapse distress, (5) An anterior sub-scale for pelvic organ prolapse distress, (6) A posterior sub-scale for pelvic organ prolapse distress, (7) An obstructive sub-scale for colorectal anal distress, (8) Incontinence, (9) Pain, and (10) A rectal prolapse sub-scale for colorectal anal distress. For each of these sub-scales, scores from from 0 to 100 (where higher scores indicate greater symptom severity). There are three additional sub-scales: (11) The urinary distress inventory, (12) The pelvic organ distress inventory, and (13) The colorectal distress inventory. Each of these ranges from 0 to 400 (with higher scores indicating greater symptom severity).
Time Frame: 12 weeks
Population: Participants who received solifenacin were asked to complete the PFDI questionnaire at 12 weeks in order to assess certain bowel, bladder, and pelvic symptoms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Solifenacin Responder | Solifenacin Non-Responder
Number analyzed (Participants) | 37 | 13
units on a scale
  Obstructive Discomfort Score | 5.77 [0 to 17.31] | 7.69 [1.92 to 26.92]
  Irritative Score | 12.50 [5.00 to 30.00] | 32.50 [7.50 to 52.50]
  Stress Score | 8.33 [0 to 27.08] | 16.67 [6.25 to 50.00]
  Urinary Distress Inventory Score | 40.19 [12.86 to 63.37] | 60.26 [23.37 to 110.87]
  General Score | 7.14 [0 to 16.07] | 14.29 [8.93 to 25.00]
  Anterior Score | 8.33 [0 to 18.75] | 8.33 [0 to 31.25]
  Posterior Score | 0 [0 to 33.33] | 16.67 [8.33 to 33.33]
  Pelvic Organ Prolapse Distress Inventory Score | 20.83 [12.20 to 58.33] | 47.62 [31.85 to 85.12]
  Obstructive Score | 0 [0 to 33.33] | 16.67 [8.33 to 33.33]
  Pain Irritation Score | 10.71 [0 to 26.79] | 10.71 [0 to 26.79]
  Rectal Prolapse | 0 [0 to 0] | 0 [0 to 0]
  Colo-Rectal-Anal Distress Inventory Score | 17.86 [7.14 to 75.48] | 42.86 [29.52 to 66.25]
  Incontinence Score | 0 [0 to 20.00] | 10.00 [0 to 22.50]
Statistical Analysis 1: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the obstructive discomfort score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in obstructive discomfort, and and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) obstructive discomfort than the other group; Test type: Superiority or Other; p = .46, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -0.74
Statistical Analysis 2: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the irritative score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in irritation, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) irritation than the other group; Test type: Superiority or Other; p = .07, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.80
Statistical Analysis 3: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the stress score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in stress, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) stress than the other group; Test type: Superiority or Other; p = .11, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.59
Statistical Analysis 4: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the urinary distress inventory score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in urinary distress, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) urinary distress than the other group; Test type: Superiority or Other; p = .09, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.69
Statistical Analysis 5: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the general score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in general pelvic floor disease severity, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) general pelvic floor disease severity than the other group; Test type: Superiority or Other; p = .09, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.68
Statistical Analysis 6: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the anterior score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in anterior pelvic floor disease severity, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) anterior pelvic floor disease severity than the other group; Test type: Superiority or Other; p = .82, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -0.23
Statistical Analysis 7: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the posterior score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in posterior pelvic floor disease severity, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) posterior pelvic floor disease severity than the other group; Test type: Superiority or Other; p = .06, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.92
Statistical Analysis 8: Comparison: Solifenacin Responder vs Solifenacin Non-Responder; For the pelvic organ prolapse distress score, the non-parametric Mann-Whitney test was used to compare the responder and non-responder groups due to low sample size in the non-responder group (n = 13). The null hypothesis is that there is no difference between the two groups in pelvic organ prolapse distress, and the two-sided alternative hypothesis is that one of the two groups has higher (or lower) pelvic organ prolapse distress than the other group; Test type: Superiority or Other; p = .07, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = -1.85

ADVERSE EVENTS:
Time Frame: Participants who received solifenacin were assessed for adverse events over 12 weeks. Control participants who did not receive solifenacin, however, were only seen at baseline (0 weeks).
Arm/Group | Urinary Urge Incontinence | Non-Urinary Urge Incontinence
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/0
Other Adverse Events (participants affected / at risk) | 10/74 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urinary Urge Incontinence (N=74) | Non-Urinary Urge Incontinence (N=0)
Dry Mouth (General disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Elevated Blood Pressure (General disorders) | 1 (1) | 0 (0)
Hives (Immune system disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No